CLINICAL TRIAL: NCT00572910
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Immunogenicity of Merck Staphylococcus Aureus Vaccine (V710) in Adult Patients With End-Stage Renal Disease on Chronic Hemodialysis
Brief Title: A Study to Evaluate the Safety and Immunogenicity of V710 in Adults With Kidney Disease on Hemodialysis (V710-005)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V710-005; 2007_609
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Results first posted 2011-08-15 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Staphylococcus Aureus Infection
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- V710 - Group 1 (Experimental): V710 (60 mcg without MAA) on Day 1 and Day 28 followed by third dose of V710 or placebo on Day 180.
  Interventions: Biological: V710 Comparator: Placebo (PBO)
- V710 - Group 2 (Experimental): V710 (60 mcg without MAA) on Day 1 and Placebo on Day 28 followed by third dose of V710 or placebo on Day 180.
  Interventions: Biological: V710 Comparator: Placebo (PBO)
- V710 - Group 3 (Experimental): V710 (60 mcg with MAA) on Day 1 and Day 28 followed by third dose of V710 or placebo on Day 180.
  Interventions: Biological: V710 Comparator: Placebo (PBO)
- V710 - Group 4 (Experimental): V710 (60 mcg with MAA) on Day 1 and Placebo on Day 28 followed by third dose of V710 or placebo on Day 180.
  Interventions: Biological: V710 Comparator: Placebo (PBO)
- V710 - Group 5 (Experimental): V710 (90 mcg with MAA) on Day 1 and Day 28 followed by third dose of V710 or placebo on Day 180.
  Interventions: Biological: V710 Comparator: Placebo (PBO)
- Group 6 (Placebo Comparator): Placebo on Day 1, 28 and 180.
  Interventions: Biological: Comparator: Placebo (PBO)

INTERVENTIONS:
Biological: Comparator: Placebo (PBO) — Group 6: Placebo (PBO / PBO / PBO)
  Arms: Group 6
Biological: V710 Comparator: Placebo (PBO) — Group 5A: V710 (90 mcg / 90 mcg / 90 mcg) with MAA
  Group 5B: V710 (90 mcg / 90 mcg / PBO) with MAA
  Arms: V710 - Group 5
Biological: V710 Comparator: Placebo (PBO) — Group 4A: V710 (60 mcg / PBO / 60 mcg) with MAA
  Group 4B: V710 (60 mcg / PBO / PBO) with MAA
  Arms: V710 - Group 4
Biological: V710 Comparator: Placebo (PBO) — Group 3A: V710 (60 mcg / 60 mcg / 60 mcg) with MAA
  Group 3B: V710 (60 mcg / 60 mcg / PBO) with MAA
  Arms: V710 - Group 3
Biological: V710 Comparator: Placebo (PBO) — Group 2A: V710 (60 mcg / PBO / 60 mcg) without MAA
  Group 2B: V710 (60 mcg / PBO / PBO) without MAA
  Arms: V710 - Group 2
Biological: V710 Comparator: Placebo (PBO) — Group 1A: V710 (60 mcg / 60 mcg / 60 mcg) without MAA
  Group 1B: V710 (60 mcg / 60 mcg / PBO) without MAA
  Arms: V710 - Group 1

SUMMARY:
This is a study to evaluate the safety and immunogenicity of V710 with and without Merck Aluminum Adjuvant (MAA) in adult participants with end-stage kidney disease who are on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with end stage kidney disease and is on hemodialysis
* Female patients who are able to have children must have a negative urine pregnancy tests

Exclusion Criteria:

* Developed a serious infection within the past 12 months; allergy to the components of the vaccine
* Has been vaccinated with a live virus within the past 30 days or are scheduled to be vaccinated with a live virus in the next 60 days
* Received V710 vaccine before

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2008-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Moustafa M, Aronoff GR, Chandran C, Hartzel JS, Smugar SS, Galphin CM, Mailloux LU, Brown E, Dinubile MJ, Kartsonis NA, Guris D. Phase IIa study of the immunogenicity and safety of the novel Staphylococcus aureus vaccine V710 in adults with end-stage renal disease receiving hemodialysis. Clin Vaccine Immunol. 2012 Sep;19(9):1509-16. doi: 10.1128/CVI.00034-12. Epub 2012 Jul 25. PMID 22837094

RESULTS

PARTICIPANT FLOW:
Groups:
- V710 (60 mcg / 60 mcg / 60 mcg): Participants in Group 1A who were vaccinated with V710 (60 mcg / 60 mcg / 60 mcg) without MAA.
- V710 (60 mcg / 60 mcg / PBO): Participants in Group 1B who were vaccinated with V710 (60 mcg / 60 mcg / PBO) without MAA.
- V710 (60 mcg / PBO / 60 mcg): Participants in Group 2A who were vaccinated with V710 (60 mcg / PBO / 60 mcg) without MAA.
- V710 (60 mcg / PBO / PBO): Participants in Group 2B who were vaccinated with V710 (60 mcg / PBO / PBO) without MAA.
- V710 (60 mcg / 60 mcg / 60 mcg) + MAA: Participants in Group 3A who were vaccinated with V710 (60 mcg / 60 mcg / 60 mcg) with MAA.
- V710 (60 mcg / 60 mcg / PBO) + MAA: Participants in Group 3B who were vaccinated with V710 (60 mcg / 60 mcg /PBO) with MAA.
- V710 (60 mcg / PBO / 60 mcg) + MAA: Participants in Group 4A who were vaccinated with V710 (60 mcg / PBO / 60 mcg) with MAA.
- V710 (60 mcg / PBO / PBO) + MAA: Participants in Group 4B who were vaccinated with V710 (60 mcg / PBO / PBO) with MAA.
- V710 (90 mcg / 90 mcg / 90 mcg) + MAA: Participants in Group 5A who were vaccinated with V710 (90 mcg / 90 mcg / 90 mcg) with MAA.
- V710 (90 mcg / 90 mcg / PBO) + MAA: Participants in Group 5B who were vaccinated with V710 (90 mcg / 90 mcg / PBO) with MAA.
- Placebo (PBO / PBO / PBO): Participants in Group 6 who were vaccinated with Placebo (PBO / PBO / PBO).
Period: Overall Study
Arm/Group | V710 (60 mcg / 60 mcg / 60 mcg) | V710 (60 mcg / 60 mcg / PBO) | V710 (60 mcg / PBO / 60 mcg) | V710 (60 mcg / PBO / PBO) | V710 (60 mcg / 60 mcg / 60 mcg) + MAA | V710 (60 mcg / 60 mcg / PBO) + MAA | V710 (60 mcg / PBO / 60 mcg) + MAA | V710 (60 mcg / PBO / PBO) + MAA | V710 (90 mcg / 90 mcg / 90 mcg) + MAA | V710 (90 mcg / 90 mcg / PBO) + MAA | Placebo (PBO / PBO / PBO)
Started | 19 | 18 | 19 | 18 | 19 | 19 | 19 | 19 | 19 | 19 | 18
Completed | 15 | 15 | 17 | 14 | 17 | 16 | 15 | 15 | 16 | 13 | 15
Not Completed | 4 | 3 | 2 | 4 | 2 | 3 | 4 | 4 | 3 | 6 | 3
Not completed — Adverse Event | 1 | 2 | 0 | 2 | 0 | 0 | 4 | 2 | 1 | 3 | 2
Not completed — Lost to Follow-up | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 1 | 0 | 1 | 3 | 0 | 2 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- V710 (60 mcg / 60 mcg): Participants who were vaccinated with V710 (60 mcg without MAA) on Day 1 and Day 28.
- V710 (60 mcg / PBO): Participants who were vaccinated with V710 (60 mcg without MAA) on Day 1 and Placebo on Day 28.
- V710 (60 mcg / 60 mcg) + MAA: Participants who were vaccinated with V710 (60 mcg with MAA) on Day 1 and Day 28.
- V710 (60 mcg / PBO) + MAA: Participants who were vaccinated with V710 (60 mcg with MAA) on Day 1 and Placebo on Day 28.
- V710 (90 mcg / 90 mcg) + MAA: Participants who were vaccinated with V710 (90 mcg with MAA) on Day 1 and Day 28.
- Placebo (PBO / PBO): Participants who were vaccinated with Placebo on Day 1 and Day 28.
- Total: Total of all reporting groups
Arm/Group | V710 (60 mcg / 60 mcg) | V710 (60 mcg / PBO) | V710 (60 mcg / 60 mcg) + MAA | V710 (60 mcg / PBO) + MAA | V710 (90 mcg / 90 mcg) + MAA | Placebo (PBO / PBO) | Total
Number analyzed (Participants) | 37 | 37 | 38 | 38 | 38 | 18 | 206
Age, Customized [Number; unit: Participants]
  <50 years of age | 10 | 14 | 14 | 5 | 14 | 6 | 63
  >=50 years of age | 27 | 23 | 24 | 33 | 24 | 12 | 143
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 19 | 14 | 16 | 7 | 84
  Male | 24 | 22 | 19 | 24 | 22 | 11 | 122

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Fold-rise (GMFR) in 0657n-specific Immunoglobulin G (IgG) Antibody Concentration From Baseline to 28 Days After the Administration of the Second V710 Vaccination
Description: Participants whose GMFR in anti-0657n IgG antibody concentration was measured by the LUMINEX™ assay from Baseline to 28 days after the administration of the second vaccination of V710 for the 3 groups receiving 2 doses of V710 (60 mcg without MAA) Group 1, (60 mcg with MAA) Group 3 and (90 mcg with MAA) Group 5.
Time Frame: Prevaccination to 56 days postvaccination
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- V710 (60 mcg Without MAA) - Group 1: Participants in Group 1 were vaccinated with V710 (60 mcg without MAA) on Day 1 and Day 28.
- V710 (60 mcg With MAA) - Group 3: Participants in Group 3 were vaccinated with V710 (60 mcg with MAA) on Day 1 and Day 28.
- V710 (90 mcg With MAA) - Group 5: Participants in Group 5 were vaccinated with V710 (90 mcg with MAA) on Day 1 and Day 28.
Arm/Group | V710 (60 mcg Without MAA) - Group 1 | V710 (60 mcg With MAA) - Group 3 | V710 (90 mcg With MAA) - Group 5
Number analyzed (Participants) | 36 | 37 | 36
Ratio | 18.9 [13.7 to 26.1] | 15.1 [11.0 to 20.8] | 17.8 [13.0 to 24.3]

2. Secondary Outcome: GMFR in 0657n-specific IgG Antibody Concentration From Baseline to Day 28 After the Administration of the First V710 Vaccination
Description: Participants whose GMFR in anti-0657n IgG antibody concentration was measured from Baseline to Day 28 for the 3 Groups receiving 1 dose of V710 (60 mcg without MAA) Group 1 and 2 combined, (60 mcg with MAA) Group 3 and 4 combined and (90 mcg with MAA) Group 5.
Time Frame: Prevaccination to 28 days postvaccination
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- V710 - Group 1 and 2: Participants in Group 1 were vaccinated with V710 (60 mcg without MAA) on Day 1 and Day 28 followed by third dose of V710 or placebo on Day 180.
  Participants Group 2 were vaccinated with V710 (60 mcg without MAA) on Day 1 and Placebo on Day 28 followed by third dose of V710 or placebo on Day 180.
- V710 - Group 3 and 4: Participants in Group 3 were vaccinated with V710 (60 mcg with MAA) on Day 1 and Day 28 followed by third dose of V710 or placebo on Day 180.
  Participants in Group 4 were vaccinated with V710 (60 mcg with MAA) on Day 1 and Placebo on Day 28 followed by third dose of V710 or placebo on Day 180.
- V710 - Group 5: Participants in Group 5 were vaccinated with V710 (90 mcg with MAA) on Day 1 and Day 28 followed by third dose of V710 or placebo on Day 180.
Arm/Group | V710 - Group 1 and 2 | V710 - Group 3 and 4 | V710 - Group 5
Number analyzed (Participants) | 73 | 74 | 36
Ratio | 11.9 (9.0) [9.0 to 15.6] | 12.9 (12.9) [9.8 to 16.9] | 12.9 [8.8 to 18.8]

3. Secondary Outcome: GMFR in 0657n-specific IgG Antibody Concentration From Baseline to Day 180 After the Administration of the First V710 Vaccination
Description: Participants whose GMFR in anti-0657n IgG antibody concentration was measured from Baseline to Day 180 for the 3 Groups receiving 2 doses of V710 28 days apart (60 mcg without MAA) Group 1, (60 mcg with MAA) Group 3 and (90 mcg with MAA) Group 5.
Time Frame: Prevaccination to 180 days postvaccination
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- V710 - Group 1: Participants in Group 1 were vaccinated V710 (60 mcg without MAA) on Day 1 and Day 28 followed by third dose of V710 or placebo on Day 180.
- V710 - Group 3: Participants in Group 2 were vaccinated V710 (60 mcg with MAA) on Day 1 and Day 28 followed by third dose of V710 or placebo on Day 180.
- V710 - Group 5: Participants in Group 5 were vaccinated V710 (90 mcg with MAA) on Day 1 and Day 28 followed by third dose of V710 or placebo on Day 180.
Arm/Group | V710 - Group 1 | V710 - Group 3 | V710 - Group 5
Number analyzed (Participants) | 36 | 37 | 36
Ratio | 8.5 [6.2 to 11.8] | 5.7 [4.2 to 7.9] | 7.6 [5.5 to 10.6]

4. Secondary Outcome: GMFR in 0657n-specific IgG Antibody Concentration From Baseline to 56 Days After the Administration of a Single V710 Vaccination
Description: Participants whose GMFR in 0657n-specific IgG antibody concentration from Baseline to Day 56 for the 2 Groups receiving a single dose of V710 (60 mcg without MAA followed by Placebo 28 Days later) Group 2, and (60 mcg with MAA followed by Placebo 28 days later) Group 4.
Time Frame: Prevaccination to 56 days postvaccination
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- V710 - Group 2: Participants in Group 2 were vaccinated V710 (60 mcg without MAA) on Day 1 and Placebo on Day 28 followed by third dose of V710 or placebo on Day 180.
- V710 - Group 4: Participants in Group 4 were vaccinated V710 (60 mcg with MAA) on Day 1 and Placebo on Day 28 followed by third dose of V710 or placebo on Day 180.
Arm/Group | V710 - Group 2 | V710 - Group 4
Number analyzed (Participants) | 37 | 37
Ratio | 9.6 [7.1 to 13.1] | 11.8 [8.6 to 16.1]

5. Secondary Outcome: GMFR in 0657n-specific IgG Antibody Concentration From Baseline as Measured at 8 Predefined Timepoints
Description: Participants whose GMFR in 0657n-specific IgG antibody concentration from baseline through Day 360 for all groups (including Days 28, 56, 84,180, 210, 270, and 360) to assess the durability and kinetics of the immune response.
Time Frame: Prevaccination to 360 days post vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- V710 (60 mcg / 60 mcg / PBO) + MAA: Participants in Group 3B who were vaccinated with V710 (60 mcg / 60 mcg / PBO) with MAA.
Arm/Group | V710 (60 mcg / 60 mcg / 60 mcg) | V710 (60 mcg / 60 mcg / PBO) | V710 (60 mcg / PBO / 60 mcg) | V710 (60 mcg / PBO / PBO) | V710 (60 mcg / 60 mcg / 60 mcg) + MAA | V710 (60 mcg / 60 mcg / PBO) + MAA | V710 (60 mcg / PBO / 60 mcg) + MAA | V710 (60 mcg / PBO / PBO) + MAA | V710 (90 mcg / 90 mcg / 90 mcg) + MAA | V710 (90 mcg / 90 mcg / PBO) + MAA | Placebo (PBO / PBO / PBO)
Number analyzed (Participants) | 18 | 18 | 19 | 18 | 19 | 18 | 19 | 18 | 17 | 19 | 18
Ratio
  Day 1 | 22.2 [13.6 to 36.4] | 19.9 [11.7 to 34.1] | 36.3 [24.3 to 54.0] | 24.6 [14.1 to 42.8] | 26.9 [16.6 to 43.8] | 33.7 [20.1 to 56.8] | 36.6 [23.6 to 56.7] | 26.6 [16.9 to 41.9] | 24.4 [15.1 to 39.3] | 25.4 [17.4 to 37.1] | 30.2 [20.7 to 44.0]
  Day 28 | 19.4 [8.0 to 47.0] | 13.4 [8.2 to 21.9] | 9.2 [5.1 to 16.6] | 9.8 [5.1 to 18.5] | 11.7 [6.5 to 21.2] | 10.8 [6.0 to 19.6] | 11.4 [6.0 to 22.0] | 14.4 [9.6 to 21.6] | 16.3 [9.2 to 28.8] | 11.4 [5.7 to 22.8] | 1.2 [0.9 to 1.5]
  Day 56 | 30.3 [17.7 to 51.9] | 14.6 [8.6 to 24.8] | 10.3 [5.9 to 18.0] | 7.8 [4.5 to 13.4] | 17.3 [10.6 to 28.3] | 12.8 [8.4 to 19.5] | 9.1 [5.3 to 15.6] | 13.1 [8.6 to 20.1] | 19.5 [11.7 to 32.6] | 17.5 [9.0 to 34.0] | 1.1 [0.9 to 1.4]
  Day 84 | 26.5 [16.2 to 43.3] | 12.1 [7.1 to 20.5] | 7.8 [4.6 to 13.1] | 6.9 [3.8 to 12.6] | 13.7 [8.7 to 21.5] | 13.0 [8.3 to 20.4] | 7.7 [4.1 to 14.3] | 10.0 [6.1 to 16.2] | 18.8 [11.4 to 30.7] | 17.2 [8.7 to 33.9] | 1.6 [0.8 to 3.0]
  Day 180 | 13.0 [7.5 to 22.6] | 7.3 [4.9 to 11.1] | 4.0 [2.4 to 6.5] | 4.2 [2.6 to 6.7] | 5.7 [2.7 to 11.9] | 5.8 [3.7 to 8.9] | 3.7 [2.3 to 6.0] | 5.5 [3.2 to 9.4] | 8.5 [5.1 to 14.1] | 10.1 [5.5 to 18.6] | 1.0 [0.8 to 1.3]
  Day 210 | 13.6 [7.8 to 23.8] | 5.6 [3.4 to 9.3] | 7.0 [4.4 to 11.0] | 4.1 [2.2 to 7.5] | 10.1 [6.3 to 16.1] | 5.4 [3.4 to 8.5] | 6.1 [4.0 to 9.2] | 4.4 [2.6 to 7.4] | 11.3 [6.6 to 19.4] | 7.7 [4.4 to 13.6] | 1.1 [0.9 to 1.3]
  Day 270 | 8.7 [5.5 to 13.6] | 4.0 [2.6 to 6.1] | 5.5 [3.5 to 8.7] | 3.6 [2.0 to 6.4] | 8.2 [5.2 to 12.8] | 3.7 [2.3 to 6.0] | 5.3 [3.6 to 7.9] | 3.9 [2.5 to 6.3] | 10.7 [5.8 to 19.9] | 5.8 [2.9 to 11.6] | 0.9 [0.5 to 1.7]
  Day 360 | 5.9 [3.9 to 8.8] | 3.4 [1.8 to 6.3] | 3.9 [2.6 to 5.8] | 3.5 [1.7 to 7.2] | 4.6 [2.6 to 8.2] | 2.9 [1.9 to 4.4] | 3.5 [2.3 to 5.2] | 3.1 [1.9 to 4.9] | 6.6 [4.0 to 11.0] | 5.2 [2.9 to 9.4] | 1.5 [0.9 to 2.4]

6. Primary Outcome: Number of Participants With Adverse Experiences (AE)/Serious Adverse Experiences (SAE)
Description: Participants with Adverse Experiences (AE) / Serious Adverse Experiences (SAE) occurring Day 1 through Day 14 following vaccinations 1, 2, and 3.
  Participants with specific SAEs including any vaccine-related SAEs, any SAEs involving a Staphylococcus aureus (S. aureus) infection, or any AEs leading to death occurring Day 1 through Day 360 following vaccination.
Time Frame: Days 1-14 following each vaccination for any AE/SAE and Days 1-360 for any vaccine-related SAEs, S. aureus SAEs, or deaths.
Measure: Number; unit: Participants
Arm/Group | V710 (60 mcg / 60 mcg / 60 mcg) | V710 (60 mcg / 60 mcg / PBO) | V710 (60 mcg / PBO / 60 mcg) | V710 (60 mcg / PBO / PBO) | V710 (60 mcg / 60 mcg / 60 mcg) + MAA | V710 (60 mcg / 60 mcg / PBO) + MAA | V710 (60 mcg / PBO / 60 mcg) + MAA | V710 (60 mcg / PBO / PBO) + MAA | V710 (90 mcg / 90 mcg / 90 mcg) + MAA | V710 (90 mcg / 90 mcg / PBO) + MAA | Placebo (PBO / PBO / PBO)
Number analyzed (Participants) | 18 | 18 | 19 | 18 | 19 | 18 | 19 | 18 | 17 | 19 | 18
Participants
  Participants with any AE's (Day 1 - 14) | 8 | 9 | 5 | 6 | 9 | 11 | 10 | 9 | 10 | 10 | 7
  Participants with any SAE's (Day 1 - 14) | 1 | 1 | 0 | 2 | 0 | 4 | 0 | 1 | 2 | 1 | 0
  Any vaccine-related SAE's (Day 1 - 360) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any SAE's with S. aureus infection (Day 1 - 360) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 1
  Any AE's involving Death (Day 1 - 360) | 1 | 2 | 0 | 2 | 0 | 0 | 4 | 1 | 1 | 3 | 2

ADVERSE EVENTS:
Time Frame: Day 1-14 following each vaccination for all AEs (non-serious or serious). Day 1-360 for specific serious AEs (vaccine-related, resulting in death, or involving a S. aureus infection).
Description: The table "Serious Adverse Events" displays serious AEs reported throughout the study duration (Days 1-360). The table "Other Adverse Events" displays AEs reported Day 1-14 following any vaccination.
Groups:
- V710 (60 mcg / PBO / 60 mcg) + MAA: Participants in Group 4A who were vaccinated with V710 (60 mcg / PBO / PBO) with MAA.
Arm/Group | V710 (60 mcg / 60 mcg / 60 mcg) | V710 (60 mcg / 60 mcg / PBO) | V710 (60 mcg / PBO / 60 mcg) | V710 (60 mcg / PBO / PBO) | V710 (60 mcg / 60 mcg / 60 mcg) + MAA | V710 (60 mcg / 60 mcg / PBO) + MAA | V710 (60 mcg / PBO / 60 mcg) + MAA | V710 (60 mcg / PBO / PBO) + MAA | V710 (90 mcg / 90 mcg / 90 mcg) + MAA | V710 (90 mcg / 90 mcg / PBO) + MAA | Placebo (PBO / PBO / PBO)
Serious Adverse Events (participants affected / at risk) | 2/18 | 3/18 | 2/19 | 5/18 | 0/19 | 5/18 | 4/19 | 2/18 | 2/17 | 5/19 | 3/18
Other Adverse Events (participants affected / at risk) | 8/18 | 9/18 | 5/19 | 4/18 | 9/19 | 10/18 | 10/19 | 8/18 | 9/17 | 10/19 | 7/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V710 (60 mcg / 60 mcg / 60 mcg) (N=18) | V710 (60 mcg / 60 mcg / PBO) (N=18) | V710 (60 mcg / PBO / 60 mcg) (N=19) | V710 (60 mcg / PBO / PBO) (N=18) | V710 (60 mcg / 60 mcg / 60 mcg) + MAA (N=19) | V710 (60 mcg / 60 mcg / PBO) + MAA (N=18) | V710 (60 mcg / PBO / 60 mcg) + MAA (N=19) | V710 (60 mcg / PBO / PBO) + MAA (N=18) | V710 (90 mcg / 90 mcg / 90 mcg) + MAA (N=17) | V710 (90 mcg / 90 mcg / PBO) + MAA (N=19) | Placebo (PBO / PBO / PBO) (N=18)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V710 (60 mcg / 60 mcg / 60 mcg) (N=18) | V710 (60 mcg / 60 mcg / PBO) (N=18) | V710 (60 mcg / PBO / 60 mcg) (N=19) | V710 (60 mcg / PBO / PBO) (N=18) | V710 (60 mcg / 60 mcg / 60 mcg) + MAA (N=19) | V710 (60 mcg / 60 mcg / PBO) + MAA (N=18) | V710 (60 mcg / PBO / 60 mcg) + MAA (N=19) | V710 (60 mcg / PBO / PBO) + MAA (N=18) | V710 (90 mcg / 90 mcg / 90 mcg) + MAA (N=17) | V710 (90 mcg / 90 mcg / PBO) + MAA (N=19) | Placebo (PBO / PBO / PBO) (N=18)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensitivity of teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device malfunction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site dryness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 3 (4) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 4 (6) | 0 (0) | 2 (2) | 2 (4) | 2 (4)
Injection site haematoma (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 5 (6) | 5 (6) | 1 (1) | 3 (4) | 8 (15) | 4 (6) | 8 (13) | 5 (5) | 5 (6) | 9 (13) | 2 (3)
Injection site paraesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Injection site swelling (General disorders) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (5) | 5 (7) | 3 (3) | 2 (2) | 3 (6) | 2 (3)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shunt thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulse absent (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Venous pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No